CLINICAL TRIAL: NCT04632277
Title: Daily Intake of Magnesium From Drinking Water in Relation to Diabetes Mellites
Brief Title: Is Mg do Improve the Glycemic Control in Patients Drink a Desalinate Water
Acronym: Mg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: The Saline Water Conversion Corporation Research Institute at Al-Jubail, KSA. (Unknown)
Responsible Party: Principal Investigator, MOHAMMED ALHARIRI, Principal Investigator, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-2019-01-407
Record Dates: First submitted 2020-09-03; First posted 2020-11-17 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus; Patients; Glucose, High Blood
Keywords: Magnesium; Diabetes mellitus; Blood samples
MeSH Terms: conditions — Diabetes Mellitus | interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): A "tap water",
  Interventions: Other: Water
- Expermental recieve low MG (Experimental): Low Mg bottle water (50mg/l)
  Interventions: Dietary Supplement: Water with low Mg
- Expermental recieve high MG (Experimental): high Mg bottle water (100 mg/l)
  Interventions: Dietary Supplement: Water with high Mg

INTERVENTIONS:
Other: Water — Participants will receive a tab water
  Arms: Placebo
Dietary Supplement: Water with low Mg — Participants will receive Low Mg bottle water (50mg/l)
  Arms: Expermental recieve low MG
Dietary Supplement: Water with high Mg — Participants will receive High Mg bottle water (100mg/l)
  Arms: Expermental recieve high MG

SUMMARY:
Background and aim:

Diabetes mellitus as a chronic disease is on rise on parallel with diseases. Magnesium (Mg) supplementation may help control glycemic response among type 2 diabetes (T2D) patients. We aim to present an overview of the possible influence of drinking water in general and mineral water in particular in improving glycemic parameters in persons with type 2 diabetes.

Method:

A randomized double blind controlled clinical trial will be conducted at the Endocrine clinic (KFHU) on 900 of patients with T2DM. All subjects participated in this study will be randomly allotted into three groups (each group N=300) to which the three waters were supplied in similar bottles marked A "tap water", B "bottle water" and C "control without any intervention".

Blood samples will be taken before and after the intervention to determine the serum concentration of magnesium, Calcium, Vit D, creatinine, FBS, serum Ca, HbA1c, fasting C-peptide levels, fasting insulin levels and insulin sensitivity. Magnesium and calcium levels in urine will be expressed as the creatinine ratio

DETAILED DESCRIPTION:
Study population and design:

A randomized double blind controlled clinical trial will be conducted at the Endocrine clinic (KFHU) on 900 of patients with T2DM. This sample size was calculated at confidence interval of 95%. for the total diabetic outpatients in Endocrine clinic at KFHU during the period October 2020-May 2021.

All subjects living in the 3 catchment areas (Dammam. Khobar and Dhahran) in the eastern province before inclusion were selected.

Intervention All subjects participated in this study will be randomly (double-blind) allotted into three groups (each group N=300) to which the three waters were supplied in similar bottles marked A "tap water", B "Low Mg bottle water (50mg/l)" and C " high Mg bottle water (100 mg/l)". These doses have been chosen according to the guideline of WHO.

All patients will be asked to consume at least one liter of water/day. When preparing coffee and tea, ordinary tap water could be used. The intervention will be lasted for lasted 3 months. None of the participants will be changed their normal dietary habits during the trial.

The mean values of all the studied parameters will be checked before starting the protocol for standardization of the protocol situp of the participants. Moreover, the diary magnesium intake will be calculated by a dietitian and all the influential factors such as, demographic factors, baseline 25(OH)D, Vit D and calcium intake, Oestrogen use and sun exposure will be controlled and monitored during the research.

Inclusion criteria:

All patients with type 2 on any diabetic treatment aged 20-85 years old with hypomagnesemia (less than 0.6 mmol/L (1.46 mg/dL).

Exclusion criteria:

Type 1 diabetic patients, pregnant women, patients who use of immunosuppressive, corticosteroids, and non-steroidal anti-inflammatory, patients who have renal dysfunction or doing dialysis,

Sampling and data collection:

All participants will be seated in air-conditioned rooms and had 10-15 min of rest before measurements were taken. After signing the consent form, the demographic and clinical data of all subjects will be record including: address, education level, smoking, age, sex; and body weight and height were measured to calculate body mass index (BMI). The average of three consecutive blood pressure readings with intervals of 5-min rest will be obtained, using an electronic sphygmomanometer. All measurements and indicators will be taken at the base line and after three months of intervention.

Blood and urine samples Blood samples will be taken before and after the intervention to determine the serum concentration of serum magnesium, Calcium, Phosphorus, Vit D, creatinine, Urea, Lipid profile, Uric acid, Liver function test, Fasting blood glucose, HbA1c, fasting C-peptide levels, fasting insulin levels and insulin sensitivity. The HOMA-IR will be calculated according to the following formulas: HOMA-IR = (glucose mg x insulin level)/405. Blood samples will be collected before and after the intervention period. A sample of urine will be collected to measure Microalbuminuria. The analysis will be performed at the central laboratory, KFHU.

Research ethics:

Ethical approved and performed under the guideline of the research ethics committee of Imam Abdulrahman Bin Faisal University, Saudi Arabia and written consent will be obtained from all subjects.

Statistical analysis:

The data was entered into an SPSS. The data analysis will be divided into two steps: Descriptive statistics and analysis of variance. The quantitative data will be represented in the form of proportions (%) and of means with standard deviations. The one-way ANOVA will be used to measure the changes between groups.

Funds details:

This project will be supported by The Saline Water Conversion Corporation Research Institute at Al-Jubail, KSA.

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 2
* On any diabetic treatment

Exclusion criteria:

* Type 1 diabetic Delete repeated word
* Pregnant women
* Patients who use of immunosuppressive, corticosteroids, and non-steroidal anti-inflammatory.
* Patients who have renal dysfunction or doing dialysis.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Magnesium (Mg). | 3 months
  Serum Mg mg/dL. Baseline and 3 months
Fasting blood glucose | 3 months
  Fasting blood glucose mg/dL. Baseline and 3 months
Insulin μIU/mL | 3 months
  Serum Insulin μIU/mL. Baseline and 3 months
HbA1c | 3 months
  HbA1c. Baseline and 3 months
Serum HDL (high-density lipoprotein) | 3 months
  Serum HDL mg/dL. Baseline and 3 months
Serum LDL (low-density lipoprotein) | 3 months
  Serum LDL mg/dL. Baseline and 3 months
Serum Triglycerides | 3 months
  Serum Triglycerides mg/dL. Baseline and 3 months
Serum Cholesterol | 3 months
  Serum Cholesterol mg/dL. Baseline and 3 months

SECONDARY OUTCOMES:
Serum Calcium | 3 months
  Ca md/dL. Baseline and 3 months
Urine Microalbumin | 3 months
  microalbuminurea (30-300 mcg/mg creatinine). Baseline and 3 months
Serum Vitamin D | 3 months
  Vit D ng/mL. Baseline and 3 months
Blood Urea mg/dL | 3 months
  Baseline and 3 months
Serum Creatinine. | 3 months
  Baseline and 3 months (mg/dL)

OTHER OUTCOMES:
Body weight | 3 months
  weight in kilograms. Baseline and 3 months
Body height | 3 months
  height in meters. Baseline and 3 months
Body mass index | 3 months
  Weight in kilograms divided by the square of height in meters. Baseline and 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Mtalhariri@Iau.Edu.Sa, Dammam
  - King Fahd Hospital of the University, Khobar

IPD SHARING:
Plan to Share IPD: Undecided
No plan to share the results

REFERENCES:
- [Background] Barbagallo M, Dominguez LJ, Galioto A, Ferlisi A, Cani C, Malfa L, Pineo A, Busardo' A, Paolisso G. Role of magnesium in insulin action, diabetes and cardio-metabolic syndrome X. Mol Aspects Med. 2003 Feb-Jun;24(1-3):39-52. doi: 10.1016/s0098-2997(02)00090-0. PMID 12537988
- [Background] Larsson SC, Wolk A. Magnesium intake and risk of type 2 diabetes: a meta-analysis. J Intern Med. 2007 Aug;262(2):208-14. doi: 10.1111/j.1365-2796.2007.01840.x. PMID 17645588
- [Result] Murakami S, Goto Y, Ito K, Hayasaka S, Kurihara S, Soga T, Tomita M, Fukuda S. The Consumption of Bicarbonate-Rich Mineral Water Improves Glycemic Control. Evid Based Complement Alternat Med. 2015;2015:824395. doi: 10.1155/2015/824395. Epub 2015 Dec 21. PMID 26798400